CLINICAL TRIAL: NCT04535427
Title: Role of L-Arginine Supplementation in the Treatment of Rheumatoid Arthritis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: L-ARG-RA
Record Dates: First submitted 2020-08-22; First posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; L-arginine
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Arginine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (Placebo Comparator): Participants in this arm will receive placebo per day.
  Interventions: Drug: Placebo
- Low dose L-arginine (Experimental): Participants in this arm will receive 9g (3g tid) L-arginine per day.
  Interventions: Drug: L-arginine
- High dose L-arginine (Experimental): Participants in this arm will receive 15g (5g tid) L-arginine per day.
  Interventions: Drug: L-arginine

INTERVENTIONS:
Drug: L-arginine — Low (3g every time, 3 times a day)or high dose (5g every time, 3 times a day) of L-arginine will be administered to the experimental groups for at least 24 weeks as an add-on treatment to the current DMARDs treatments for rheumatoid arthritis.
  Arms: High dose L-arginine; Low dose L-arginine
Drug: Placebo — Placebo will be administered to the control group for at least 24 weeks as an add-on treatment to the current DMARDs treatments for rheumatoid arthritis.
  Arms: Control

SUMMARY:
To investigate the role of L-arginine supplementation in the treatment of DMARDs-refractory moderate to severe rheumatoid arthritis

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for inclusion in this study, subjects must meet all of the following criteria:

* Chinese RA patients who are between 18 and 45 years old (inclusive) when signing the consent form, with a body mass index between 19 and 29 kg/m2 (inclusive), and weigh between 60 and 90 kg.
* The subject must be diagnosed with RA, and the judgment standard meets the 2010 American College of Rheumatology (ACR)/European Alliance Against Rheumatism (EULAR) RA classification standard;
* Active RA is defined as having ≥ 6 swollen joints and ≥ 6 tender joints at screening and baseline (based on 66/68 joints, excluding distal interphalangeal joints), and at least one of the following conditions occurs during screening: ESR ≥ 28 mm/hr, or serum CRP> 10 mg/L;
* Positive rheumatoid factor or anti-cyclic citrulline peptide (CCP) during screening;
* Before using the study drug, the subject must have used MTX continuously for ≥ 12 weeks and have been stable for at least 8 weeks.
* 10-15mg/week dose and willing to use a stable dose throughout the study;
* Patients with moderate to severe disease activity after the current treatment of DMARDs, DAS28-ESR/CRP>3.2;
* Subjects taking oral corticosteroids (≤ 10 mg of prednisone or equivalent) should use a stable dose for ≥ 4 weeks before screening;
* If subjects are taking non-steroidal anti-inflammatory drugs (NSAIDs) or low-efficiency analgesics, such as tramadol, neuronal cell compounds, they must use a stable dose for ≥ 2 weeks before screening.
* Considered as eligible subjects based on the following tuberculosis screening criteria:

  1. The subject has no history of latent or active tuberculosis before screening,
  2. No signs or symptoms of active tuberculosis in the history and/or physical examination,
  3. Have not had close contact with patients with active tuberculosis recently,
  4. One chest radiograph (including anteroposterior and lateral views) taken within three months before the administration of the study drug, and qualified radiologists have confirmed that there are no active tuberculosis foci or old inactivated tuberculosis foci.
* Non-smokers, or agree to smoke no more than 10 cigarettes or no more than 2 cigars per day during the entire study period. Note: According to the rules and regulations of the research center, smoking may be prohibited during hospitalization;
* Agree to abstain from alcohol within 48 hours before the administration of the study drug and during the study hospitalization, and agree to drink no more than 10g of alcohol per day during the rest of the study;
* Agree to limit caffeine intake, with a daily limit of five cups of tea, or three cups of coffee or six cans of cola. Do not take caffeine within 4 hours before receiving the electrocardiogram;
* Agree to fully use birth control measures to prevent pregnancy (such as birth control pills, uterine contraceptive devices, or protective measures using spermicides) for at least six months after receiving study drug treatment;
* Except for taking acetaminophen and previously taken multivitamins at the recommended dose, as well as the drugs approved by the investigator and medical monitor, the subject agreed to not use prescription drugs for 14 days before receiving the study drug treatment until the end of the study , Over-the-counter medicines, herbal medicines, proprietary Chinese medicines or "natural" medicines;
* Demonstrate a clear understanding of the research and sign an informed consent (ICF);
* Personal willingness and ability to comply with the study follow-up schedule and other requirements of the study protocol.

Exclusion Criteria:

Subjects who meet any of the following criteria should not be selected for this study:

* RA patients combined with hypotension.
* RA patients combined with renal tubular acidosis and electrolyte imbalance.
* RA patients with significant gastrointestinal symptoms.
* According to the judgment of the main investigator, the subject is in a latent physical or psycho-medical state and will not be able to complete the study.
* Have had major surgery or traumatic surgery within 12 weeks before screening.
* Have received an organ transplant (except for corneal transplantation for more than three months before administration).
* Donated blood within 56 days before screening (the blood donation volume is not less than 500 mL).
* Currently suffering from malignant tumors or a history of malignant tumors.
* A history of known lymphoproliferative diseases, including lymphoma or possible signs and symptoms of lymphoproliferative diseases, such as lymphadenopathy and/or splenomegaly.
* Have a recent history of alcohol or drug abuse (within the previous 6 months).
* Positive urine toxicology screening for drugs of abuse include: cocaine, cannabidiol, phencyclidine, amphetamine, methamphetamine, benzodiazepines, barbiturates, opioids, and C Oxyphene, methaqualone, methadone and tricyclic antidepressants.
* When admitted to the research center before the study drug was administered, the urine alcohol screening or breath alcohol test results were positive.
* Have a history of latent or active granulomatous infection before screening, including histoplasmosis or coccidioidomycosis.
* Have a history of known or suspected intolerance or hypersensitivity to any biological drug treatment.
* Chest x-ray pictures taken within 3 months before the first administration of the study drug showed abnormalities suggesting malignant tumors or current active infections (including TB).
* Have nontuberculous mycobacteria or opportunistic infections (such as cytomegalovirus, pneumocystis disease, aspergillosis) within 6 months before screening.
* Have or have had a serious infection (such as sepsis, pneumonia, or pyelonephritis) or were hospitalized for infection or received fourth-generation antibiotic treatment within 2 months before screening.
* A history of chronic or recurrent infectious diseases, including but not limited to the following diseases: chronic kidney infection, chronic chest infection (for example, bronchiectasis), recurrent urinary tract infection (recurrent pyelonephritis or chronic non-dilated bladder) Inflammation), or open, draining or infectious skin wounds or ulcers.
* Serum was positive for HIV-1 or HIV-2, hepatitis B virus (HBV) or hepatitis C virus (HCV) during screening.
* Syphilis (Treponema pallidum) test (qualitative test) was positive at screening.
* The staff of the main researcher or research center and directly participate in the research or other research of the main researcher or research center, including the staff or the family members of the main researcher.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The response rate of ACR20 after 24 weeks of L-arginine administration | Week 0+3+6+9+12+15+18+21+24+26
  According to the American College of Rheumatology 20/50/70 criteria, the ACR20 is a composite measure defined as both improvement of 20% in the number of tender and number of swollen joints, and a 20% improvement in three of the following five criteria: patient global assessment, physician global assessment, functional ability measure [most often Health Assessment Questionnaire (HAQ)], visual analog pain scale, and erythrocyte sedimentation rate or C-reactive protein (CRP).The reduction ratio of ACR20 after 24 weeks of high or low dose of L-arginine or placebo administration will be observed and documented as the measurement of primary outcome.

SECONDARY OUTCOMES:
The response rate of ACR50/70 after 24 weeks of L-arginine administration | Week 0+3+6+9+12+15+18+21+24+26
  According to the American College of Rheumatology 20/50/70 criteria, ACR50/70 are the same instruments with improvement levels defined as 50% and 70% respectively versus 20% for ACR20. The reduction ratio of ACR 50/70 after 24 weeks of high or low dose of L-arginine or placebo administration will be observed and documented as the measurement of secondary outcome.
The change of DAS28/ESR | Week 0+3+6+9+12+15+18+21+24+26
  The DAS28 Scores indicate how active a patient's rheumatoid arthritis is currently, and can be trended over time. DAS stands for 'disease activity score' and the number 28 refers to the 28 joints that are examined in this assessment. The EULAR Response Criteria also allows clinicians to use DAS28 to categorize the effectiveness of a particular therapy.The formula for DAS28/ESR is (0.56*√(Tender Joint Count)+0.28*√(Swollen Joint Count)+0.7*ln(ESR)+0.014*(global health)). In this study, the change of DAS28/ESR will also be observed and documented as the measurement of secondary outcome.
Numbers of participants with treatment-related adverse events | Week 0+3+6+9+12+15+18+21+24+26
  The adverse events in each group will be observed and documented during the whole procedure to show the safety of L-arginine treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxiang Chen, PhD, Principal Investigator — Department of Rheumatology, Renji Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Department of Rheumatology, Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China

REFERENCES:
- [Background] Hannemann N, Cao S, Eriksson D, Schnelzer A, Jordan J, Eberhardt M, Schleicher U, Rech J, Ramming A, Uebe S, Ekici A, Canete JD, Chen X, Bauerle T, Vera J, Bogdan C, Schett G, Bozec A. Transcription factor Fra-1 targets arginase-1 to enhance macrophage-mediated inflammation in arthritis. J Clin Invest. 2019 Apr 16;129(7):2669-2684. doi: 10.1172/JCI96832. PMID 30990796